CLINICAL TRIAL: NCT00979459
Title: A Single Dose Study to Compare the Pharmacokinetics of Two Probe Formulations of MK-1006
Brief Title: A Study of the Pharmacokinetics of Two Formulations of MK-1006 (MK-1006-010 AM1)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1006-010; 2009_663
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-1006 80 mg DFC (Experimental): Participants received a single dose of four 20 mg dry filled capsules of MK-1006
  Interventions: Drug: MK-1006 DFC
- MK-1006 80 mg FCT (Experimental): Participants received a single dose of two 40 mg film coated tablets of MK-1006
  Interventions: Drug: MK-1006 FCT

INTERVENTIONS:
Drug: MK-1006 DFC — Each dry filled capsule contains 20 mg MK-1006
  Arms: MK-1006 80 mg DFC
Drug: MK-1006 FCT — Each film coated tablet contains 40 mg of MK-1006
  Arms: MK-1006 80 mg FCT

SUMMARY:
This study will assess the pharmacokinetics of two formulations of MK-1006. The primary hypothesis of this study is that the MK-1006 area under the curve (0 to infinity) and maximum concentration after administration of a single 80 mg dose of the dry filled capsule (DFC) and film coated tablet (FCT) formulations of MK-1006 will be similar.

ELIGIBILITY:
Inclusion Criteria:

* is a male or a female of non-child bearing potential
* has type 2 diabetes (T2D) and is either being treated with diet and exercise alone or with a single or combination oral anti-hyperglycemic agent(s)
* has been a nonsmoker for at least 6 months

Exclusion Criteria:

* has a history of stroke, chronic seizures, or major neurological disorder
* has a history of major endocrine (except T2D), gastrointestinal, cardiovascular, blood, liver, immune, kidney, respiratory, or genitourinary abnormalities or diseases
* has a history of cancer, except certain skin or cervical cancers or cancer that was successfully treated more than 10 years prior to screening
* has unstable or rapidly progressing diabetic retinopathy and/or neuropathy
* has had an eye infection or other inflammation of the eye in the 2 weeks prior to screening
* has glaucoma or is blind
* has had incisional eye surgery in the last 6 months or laser eye surgery in the last 3 months (Lasik is permitted)
* has a history of type 1 diabetes
* has symptomatic coronary artery disease
* consumes excessive amounts of alcohol and/or caffeine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-1006 DFC, Then MK-1006 FCT: Participants received a single dose of four 20 mg MK-1006 dry filled capsules (DFC) followed by a single dose of two 40 mg MK-1006 film coated tablets (FCT) after a 7 day washout period.
- MK-1006 FCT, Then MK-1006 DFC: Participants received a single dose of two 40 mg film coated tablets (FCT) of MK-1006 followed by a single dose of four 20 mg MK-1006 dry filled capsules (DFC) after a 7 day washout period.
Period: First Intervention
Arm/Group | MK-1006 DFC, Then MK-1006 FCT | MK-1006 FCT, Then MK-1006 DFC
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: 7-day Washout Period
Arm/Group | MK-1006 DFC, Then MK-1006 FCT | MK-1006 FCT, Then MK-1006 DFC
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | MK-1006 DFC, Then MK-1006 FCT | MK-1006 FCT, Then MK-1006 DFC
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Includes participants who were randomized to receive either a single dose of four 20 mg MK-1006 DFC followed by a single dose of two 40 mg MK-1006 FCT or a single dose of four 20 mg MK-1006 FCT followed by a single dose of two 40 mg MK-1006 DFC
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  <35 years | 0
  Between 35 and 65 years | 12
  >65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC(0-infinity)) for MK-1006
Description: AUC (0-infinity) is the area under the curve for the plot showing plasma concentration against time from time zero to the time of the last quantifiable concentration for two formulations of MK-1006, FCT and DFC
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96 and 120 hours post-dose
Measure: Geometric Mean (95% Confidence Interval); unit: nM*hr
Groups:
- MK-1006 80 mg FCT: Participants received a single dose of two MK-1006 40 mg FCT
- MK-1006 80 mg DFC: Participants received a single dose of four MK-1006 20 mg DFC
Arm/Group | MK-1006 80 mg FCT | MK-1006 80 mg DFC
Number analyzed (Participants) | 12 | 12
nM*hr | 5171 [4350 to 6147] | 5588 [4593 to 6798]
Statistical Analysis 1: Comparison: MK-1006 80 mg FCT vs MK-1006 80 mg DFC; Test type: Non-Inferiority or Equivalence — Administration of a single dose of two 40 mg MK-1006 FCT is similar to a single dose of four 20 mg MK-1006 DFC will be satisfied if the 90% confidence interval for the AUC(0 to infinity) geometric mean ratio (FCT/DCF) is contained within (0.70, 1.43); Geometric mean ratio = 0.93, 90% CI 2-sided [0.86 to 0.99]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for MK-1006
Description: Maximum plasma concentration for 2 formulations of MK-1006, FCT and DFC
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96 and 120 hours post-dose
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | MK-1006 80 mg FCT | MK-1006 80 mg DFC
Number analyzed (Participants) | 12 | 12
nM | 554 [429 to 715] | 519 [405 to 664]
Statistical Analysis 1: Comparison: MK-1006 80 mg FCT vs MK-1006 80 mg DFC; Test type: Non-Inferiority or Equivalence — Administration of a single dose of two 40 mg MK-1006 FCT is similar to a single dose of four 20 mg MK-1006 DFC will be satisfied if the 90% confidence interval for the Cmax geometric mean ratio (FCT/DCF) is contained within (0.70, 1.43); Geometric mean ratio = 1.07, 90% CI 2-sided [0.92 to 1.24]

3. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Time Frame: Through 30 days post-dose
Population: All participants received both formulations of MK-1006, FCT and DFC, and appear in both treatment groups.
Measure: Number; unit: participants
Groups:
- MK-1006 80 mg FCT: Participants received a single dose of two MK-1006 40 mg film coated tablets
- MK-1006 80 mg DFC: Participants received a single dose of four MK-1006 20 mg dry filled capsules
Arm/Group | MK-1006 80 mg FCT | MK-1006 80 mg DFC
Number analyzed (Participants) | 12 | 12
participants | 7 | 6

4. Secondary Outcome: Number of Participants Who Discontinued Study Medication Due to an Adverse Event
Time Frame: up to 8 days
Population: All participants received both formulations of MK-1006, FCT and DFC, and appear in both treatment groups.
Measure: Number; unit: participants
Arm/Group | MK-1006 80 mg FCT | MK-1006 80 mg DFC
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | MK-1006 80 mg FCT | MK-1006 80 mg DFC
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-1006 80 mg FCT (N=12) | MK-1006 80 mg DFC (N=12)
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Infusion Site Haematoma (General disorders) | 0 | 1
Infusion Site Inflammation (General disorders) | 0 | 1
Infusion Site Pain (General disorders) | 0 | 1
Vessel Puncture Site Haematoma (General disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.